CLINICAL TRIAL: NCT01771445
Title: Role of Interleukin-1 in the Regulation of Muscle Derived Interleukin-6 During Exercise
Acronym: MUSIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Y.Donath (Other)
Responsible Party: Sponsor-Investigator, Marc Y.Donath, Prof., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MUSIL 294/10
Record Dates: First submitted 2012-02-29; First posted 2013-01-18 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
Keywords: IL-1; IL-6; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- IL-1Ra (Active Comparator)
  Interventions: Drug: IL-1Ra
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IL-1Ra — 100mg, s.c, once only
  Arms: IL-1Ra
Drug: Placebo — 100mg, s.c., once only
  Arms: Placebo

SUMMARY:
Aim: Evaluate the regulation of muscle derived Interleukin-6 (IL-6)during exercise and in particular whether it is regulated by the Interleukin-1 (IL-1) system.

Rationale: It has been shown that IL-1 antagonism improves glycemia and insulin secretion in patients with type 2 Diabetes. However, IL-1 antagonism also decreases IL-6 levels. The effect if IL-6 on the glucose metabolism has been unclear in the past and subject to intense debate, with recent evidence indicating a beneficial role in regulating glucose metabolism. However little is known about regulation of muscle-induced IL-6 produced during exercise. It is therefore our aim to investigate whether exercise induced increases in IL-6 are dependent on the IL-1 system. If IL-1 antagonism does decrease IL-6 and along with it, the beneficial potential of IL-6, this may require additional medication like IL-6 substitution or dipeptidyl peptidase-IV (DPP-IV)antagonists.

In addition, the investigators will assess the effect of IL-1 antagonism on insulin and Glucagon like peptide-1 (GLP-1) secretion as well as muscle soreness,fatigue and vascular function in response to an acute exercise bout.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled, double blind, cross-over, proof-of-concept study.

The study will consist of one screening visit followed by 3 study visits. During the first two study visits, the subjects (20 apparently healthy, lean men) will perform a submaximal exercise bout on a treadmill for 60 minutes. Subjects will be randomly assigned into two groups consisting each of 10 subjects receiving study medication in a double-blinded, crossed over manner.

ELIGIBILITY:
Inclusion Criteria:

* male
* non-smoking
* apparently healthy
* BMI > 18 and < 26kg/m2
* Age 20-50 years
* Regular exercise including a minimum of two runs weekly of a total duration of > 2h
* Willingness to use contraceptive measures adequate to prevent the subject's partner from becoming pregnant during the study. Adequate contraceptive measures include hormonal methods used for two or more cycles prior to Screening (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), double barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, and condom used in conjunction with contraceptive foam or jelly), intrauterine methods (IUD), sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner), and abstinence.

Exclusion Criteria:

* Clinical signs of infection in the week before inclusion or history of infection during the last 3 months (CRP > 5mg/L)
* Impaired fasting glucose (fasting plasma glucose > 5.5mmol/L)
* Hematologic disease (leukocyte count < 1.5x109/L, hemoglobin < 11 g/dL, platelets < 100 x 103/uL)
* Kidney disease (creatinine > 1.5 mg/dL for men and 1.4mg/dL for woman)
* Liver disease (transaminases > 2x upper normal range)
* Heart disease
* Pulmonary disease
* Inflammatory disease
* History of carcinoma
* History of tuberculosis
* Alcohol consumption > 40g/d
* Known allergy to Kineret
* Current treatment with any drug in the week before inclusion, including vitamin supplementation (especially vitamin C and E)
* Use of any investigational drug within 30 days prior to enrollment or within 5 half-lives of the investigational drug, whichever is longer
* Subject refusing or unable to give written informed consent

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
IL6 | Change of IL6 during exercise stimulation at baseline compared to change of IL6 during exercise stimulation at day 7

SECONDARY OUTCOMES:
change of inflammatory markers (CRP, Tumor Necrosis Factor alpha, IL-1Ra) | Change of inflammatory markers during exercise stimulation at baseline compared to change of inflammatory markers during exercise stimulation at day 7
Muscle soreness | Change in muscle soreness before and after exercise stimulation at baseline compared to change in muscle soreness before and after exercise stimulation at day 7
Activity induced Fatigue (ACTIF) Scale | Change in ACTIF before and after exercise stimulation at baseline compared to change in ACTIF before and after exercise stimulation at day 7
Depression | Change in depression during exercise stimulation at baseline compared to change in depression at day 7
Change of vascular function (CAVI, pulse wave velocity, AVR) | Change in vascular function during exercise stimulation at baseline compared to change of vascular function at day 7
glucose metabolism | Change glucose metabolism during exercise stimulation at basleine compared to change in glucose metabolism during exercise stimulation at day 7
Cognition | Change in cognition during exercise stimulation at baseline compared to change in cognition at day 7
Motor strength | Change in motor strength during exercise stimulation at baseline compared to change in motor stength at day 7
Insulin | Change in insulin during exercise stimulation at baseline compared to change in insulin at day 7
Glucagon | Change in glucagon during exercise stimulation at baseline compared to change in glucagon at day 7
GLP-1 | Change in GLP-1 during exercise stimulation at baseline compared to change in GLP-1 at day 7
Cortisol | Change in cortisol during exercise stimulation at baseline compared to change in cortisol at day 7
Creatinkinase | Change in creatinkinase during exercise stimulation at baseline compared to change in creatinkinase at day 7
Growth hormone | Change of growth hormone during exercise stimulation at baseline compared to change of growth hormone during exercise stimulation at day 7
Copeptin | Change of copeptin during exercise stimulation at baseline compared to change of copeptin during exercise stimulation at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, MD, Principal Investigator — University of Basel
Locations (1):
- University Hospital of Basel, Division of Endocrinology, Basel, Basel, Switzerland

REFERENCES:
- [Derived] Nordmann TM, Seelig E, Timper K, Cordes M, Coslovsky M, Hanssen H, Schmidt-Trucksass A, Donath MY. Muscle-Derived IL-6 Is Not Regulated by IL-1 during Exercise. A Double Blind, Placebo-Controlled, Randomized Crossover Study. PLoS One. 2015 Oct 8;10(10):e0139662. doi: 10.1371/journal.pone.0139662. eCollection 2015. PMID 26448147